CLINICAL TRIAL: NCT03093649
Title: Measuring Patient-Reported Adverse Events in Oncology Practice Improves Quality of Life in Patients With Nasopharyngeal Carcinoma Undergoing Intensity Modulated Radiation Therapy: A Randomised Controlled Trial
Brief Title: Measuring Patient-Reported Adverse Events in Oncology Practice Improves Quality of Life in Nasopharyngeal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ying Sun, principal investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-FXY-003-放疗科
Record Dates: First submitted 2017-03-16; First posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient reported group (Experimental): Patients reported adverse events using patient reported outcomes version of common terminology criteria for adverse events (PRO-CTCAE) through Application (APP) during the treatment. The summary report was transferred to their clinician immediately. Oncologists would be alarmed if patients reports exceeding the pre-defined threshold.
  Interventions: Other: adverse events using patient-reported outcomes version of common terminology criteria for adverse events (PRO-CTCAE) questionaire
- non-reported group (Active Comparator): Patients in this group received normal care during the treatment without completing patient reported outcomes version of common terminology criteria for adverse events (PRO-CTCAE)
  Interventions: Other: do not report adverse events through patient-reported outcomes version of common terminology criteria for adverse events (PRO-CTCAE) questionaire

INTERVENTIONS:
Other: adverse events using patient-reported outcomes version of common terminology criteria for adverse events (PRO-CTCAE) questionaire — The intervention was administrated through APP
  Arms: patient reported group
Other: do not report adverse events through patient-reported outcomes version of common terminology criteria for adverse events (PRO-CTCAE) questionaire — patients receive normal care and visit
  Arms: non-reported group

SUMMARY:
Although patient-reported adverse events have been promoted as an essential element in clinical trials and daily managements, their efficacy remained unknown. The purpose of this trial was to determine the effect of the patient-reported adverse events during the treatment on the improvements on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing carcinoma (according to WHO histological type)
* No evidence of distant metastasis (M0)
* Performance status: PS 0~2
* Receive standard treatment
* Able to read and understand the questionnaires
* Not exhibiting overt psychopathology
* Willing to give feedback to physicians and written informed consent was obtained

Exclusion Criteria:

* WHO type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Treatment with palliative intent.
* Prior malignancy (except adequately treated carcinoma in-situ of the cervix or basal/squamous cell carcinoma of the skin)
* Previous chemotherapy or radiotherapy (except non-melanomatous skin cancers outside the intended RT treatment volume)
* Patient is pregnant or lactating
* Severe intercurrent disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Score of physical functioning in quality of life | within 1 week of study completion
  Score of physical functioning in quality of life

SECONDARY OUTCOMES:
3-year overall survival | 3 year after diagnosis
  overall survival at three year after diagnosis
3-year progression-free survival | 3 year after diagnosis
  progression-free survival at three year after diagnosis
3-year local-regional free survival | 3 year after diagnosis
  local-regional free survival at three year after diagnosis
3-year metastatic-free survival | 3 year after diagnosis
  metastatic-free survival at three year after diagnosis
completion rate | within 1 week of study completion
  completion rate
degrees of patients satisfaction regarding the treatment process | within 1 week of study completion
  degrees of patients satisfaction regarding the treatment process
response rate | 1 month after study completion
  response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China